CLINICAL TRIAL: NCT05484752
Title: Efficacy of Peripheral Magnetic Stimulation to Reduce Pain in Knee Osteoarthritis: A Randomized Controlled Trial.
Brief Title: Efficacy of Peripheral Magnetic Stimulation to Reduce Pain in Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ApiphanRama
Record Dates: First submitted 2022-08-01; First posted 2022-08-02 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repetitive Peripheral Magnetic Stimulation (Experimental): Repetitive Peripheral Magnetic Stimulation 1 session
  Interventions: Device: Repetitive Peripheral Magnetic Stimulation; Behavioral: Education
- Sham Repetitive Peripheral Magnetic Stimulation (Sham Comparator): Sham Repetitive Peripheral Magnetic Stimulation 1 session
  Interventions: Behavioral: Education

INTERVENTIONS:
Device: Repetitive Peripheral Magnetic Stimulation — Repetitive Peripheral Magnetic Stimulation at knee joint 1 session
  Arms: Repetitive Peripheral Magnetic Stimulation
Behavioral: Education — Conventional exercise and life style modification

SUMMARY:
To investigate effects of repetitive peripheral magnetic stimulation (PMS) on pain reduction in knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Primary knee osteoarthritis patients who have had knee pain for at least 6 months and age more than 50 years, had morning stiffness not more than 30 minutes or crepitation.
* Kellgren and Lawrence classification 2-4
* Visual analog scale of pain 4 or higher.

Exclusion Criteria:

* Patients with other musculoskeletal problems associated with knee joint
* Patient with history of physical therapy in past 1 month
* Patient with pacemaker, cochlear implant or cerebral shunt
* Patient with history of knee surgery
* Patient with neurological or other severe disease
* Patient with previous seizure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change of Visual analog scale | Change from baseline Visual analog scale at immediately after intervention and Change from Baseline visual analog scale at 1 week.
  Pain measurement Score from 0-10, 0 means no pain and 10 means maximum pain. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Modified Western Ontario and McMaster University Osteoarthritis Index | Change from Baseline Modified Western Ontario and McMaster University Osteoarthritis Index at 1 week.
  To assessing pain, stiffness, and function in patients with osteoarthritis. Score from 0-220. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Apiphan Iamchaimongkol, M.D., Study Director — Ramathibodi Hospital
Locations (1):
- Physical medicine and rehabilitation, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pujol J, Pascual-Leone A, Dolz C, Delgado E, Dolz JL, Aldoma J. The effect of repetitive magnetic stimulation on localized musculoskeletal pain. Neuroreport. 1998 Jun 1;9(8):1745-8. doi: 10.1097/00001756-199806010-00014. PMID 9665594
- See also: The effect of repetitive magnetic stimulation on localized musculoskeletal pain. — http://doi.org/10.1097/00001756-199806010-00014